CLINICAL TRIAL: NCT02262572
Title: Relative Bioavailability of Telmisartan and HCTZ p.o. (80 mg Telmisartan/12.5 mg HCTZ) in Two Experimental Formulations (Given t.i.d. for One Day Each) Compared to the Standard Formulation 80 mg Telmisartan/12.5 mg HCTZ (MicardisPlus®), Given t.i.d. for One Day in Healthy Female and Male Subjects. A Three-way Crossover, Open, Randomised Study
Brief Title: Relative Bioavailability of Telmisartan and HCTZ in Two Experimental Formulations Compared to the Standard Formulation Telmisartan and HCTZ in Healthy Female and Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.415
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; telmisartan, hydrochlorothiazide drug combination

ARMS (3):
- Telmisartan /HCTZ - compression tablet (DC) (Experimental)
  Interventions: Drug: Telmisartan /HCTZ - compression tablet (DC)
- Telmisartan /HCTZ - dry granulation tablet (DG) (Experimental)
  Interventions: Drug: Telmisartan /HCTZ - dry granulation tablet (DG)
- Telmisartan /HCTZ - present commercial formulation (Active Comparator)
  Interventions: Drug: Telmisartan /HCTZ - present commercial formulation

INTERVENTIONS:
Drug: Telmisartan /HCTZ - compression tablet (DC)
  Arms: Telmisartan /HCTZ - compression tablet (DC)
Drug: Telmisartan /HCTZ - dry granulation tablet (DG)
  Arms: Telmisartan /HCTZ - dry granulation tablet (DG)
Drug: Telmisartan /HCTZ - present commercial formulation
  Other Names: MicardisPlus®
  Arms: Telmisartan /HCTZ - present commercial formulation

SUMMARY:
Study to assess the comparative pharmacokinetics of telmisartan/HCTZ in two new formulations based on sodium salt compared to the present commercial formulation (MicardisPlus®)

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following criteria will be eligible for participation in the study:

* Healthy male and female subjects according to the following criteria: based upon a complete medical history, including the physical examination, vital signs (BP, HR), 12-lead ECG, clinical laboratory tests.
* Laboratory values within a clinically defined reference range
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Age >=18 and Age <=55 years
* Body mass index (BMI) >=18.5 and <=29.9 kg/m2
* Able to communicate well with the investigator and to comply with study requirements
* Good condition of veins

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, heart rate, and electrocardiogram) deviating from normal and of clinical relevance
* Supine blood pressure at screening of systolic ≤ 110 mm Hg and diastolic ≤ 60 mmHg
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of an allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of any drugs, which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (more than 10 cigarettes or three cigars or three pipes/day)
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation or loss of more than 400 mL within four weeks prior to administration or during the trial
* Excessive physical activities (within five days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* History of hereditary fructose intolerance
* Veins unsuited for i.v. puncture on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture, etc.)
* Inability to comply with the dietary regimen of study centre
* Inability to comply with the investigator's instructions.

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. oral contraceptives, sterilization, intrauterine device (IUD)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-04; Primary Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after drug administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
Amount of HCTZ excreted in urine over 48 hours (%Ae0-48h) | up to 48 hours after drug administration

SECONDARY OUTCOMES:
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 72 hours after drug administration
t1/2 (Terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
CLtot/F (Apparent clearance of the analyte in plasma following extravascular administration) | up to 72 hours after drug administration
MRTtot (Total mean residence time) | up to 72 hours after drug administration
Vz/F (Apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours after drug administration
Number of subjects with adverse events | up to 32 days
Number of subjects with clinically significant findings in vital signs | up to 32 days
  blood pressure, pulse rate
Number of subjects with clinically significant findings in 12 lead ECG | up to 32 days
Investigator's assessment of tolerability on a 4-point scale | up to 32 days